CLINICAL TRIAL: NCT03025152
Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Spleen Qi Deficiency and Radical Gastrectomy for Gastric Cancer: A Multicenter, Randomized, Double-blinded, Parallel-group, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Spleen Qi Deficiency and Radical Gastrectomy for Gastric Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High attrition rate up to 37.7% at one year's follow-up
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xu Zhou, Principal Investigator, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JXUTCM-EBM-02
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer; Gastrointestinal Disease
Keywords: Hou Gu Mi Xi; Shen Ling Bai Zhu San; radical gastrectomy; gastric cancer; traditional Chinese medicine; randomized controlled trial
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hou Gu Mi Xi (Experimental): Patients in this arm receive Hou Gu Mi Xi, with an oral dose of 10 g/day during entire follow up period (2 years).
  Interventions: Dietary Supplement: Hou Gu Mi Xi
- placebo (Placebo Comparator): Patients in this arm receive placebo, with an oral dose of 10 g/day during entire follow up period (2 years).
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Hou Gu Mi Xi — Hou Gu Mi Xi is a dietary therapy form of Shen Ling Bai Zhu San, which removes atractylodes and platycodon grandiflorum, adds perilla leaf for adapting a dietary therapy.
  Arms: Hou Gu Mi Xi
Other: placebo — The placebo has same appearance, taste and smell as Hou Gu Mi Xi.
  Arms: placebo

SUMMARY:
This trial aims to determine whether Hou Gu Mi Xi is an effective treatment for improving symptoms and indicators in patients with spleen qi deficiency and radical gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
The incidence of gastric cancer ranks high in many countries around the world. Although along with the development of economy and medical condition the incidence of gastric cancer appears a trend of decrease in developed countries, it is still one of most common cancers in Asia. There are more new gastric cancer cases in China compared with other countries every year. According to an epidemiological survey by World Health Organization, 5-year prevalence of gastric cancer was 53.7/10,000 in China - it is only lower than Japan. For the early gastric cancer, radical gastrectomy, is the most important treatment, which could significantly prolong disease-free survival and overall survival. However, the severe damage of surgery and following radiation and chemotherapy in intestinal tract usually leads patients to be a constitution of spleen qi deficiency, a concept of traditional Chinese medicine (TCM) that mainly involves digestive symptoms, such as poor appetite, abnormal stool (loose, diarrhea) and abdominal distention. Therefore, how to resolve and protect the function of intestinal tract, and change the constitution of spleen qi deficiency postoperatively is important for improving quality of life and reducing the recurrence rate of cancer.

Shen Ling Bai Zhu San, a classic Chinese medicinal formulae originally described in Tai Ping Hui Min He Ji Ju Fang in the Song Dynasty (1102 AD), is composed of ginseng, tuckahoe, atractylodes, baked licorice, coixenolide, Chinese yam, lotus seed, shrinkage fructus amomi, platycodon grandiflorum, white hyacinth bean, and dried orange peel. It has effects of replenishing qi and invigorating spleen (spleen is a TCM conception that differs from western medicine), as well as penetrating wet and antidiarrheal. It is mainly used for treating the syndrome of spleen qi deficiency, including dyspepsia, chest and stomach distress, borborygmus and diarrhea, limb weakness, thin body, sallow complexion, pale tongue with white and greasy coating, and weak and slow pulse, etc. In the theory of TCM, spleen is the source for producing qi and blood and thus is the root of life. Shen Ling Bai Zhu San could invigorate spleen by supplying spleen and remove wet, and finally nourish the stomach and intestine. Previous pharmacologic studies also revealed that Shen Ling Bai Zhu San could adjust function of anaerobic and aerobic bacteria in gastrointestinal tract; specifically, it could improve the proliferation of probiotics (such as bifidobacterium) and inhibit the main resistance strains (such as enterococcus) and thus has an effect to improve gastrointestinal symptoms.

According to the experience of TCM, the constitution of patients who are undergoing radiation and chemotherapy is usually yin deficiency, but changes to spleen qi deficiency due to digestive disorders after those treatment. Therefore, Shen Ling Bai Zhu San is expected to improve symptoms in patients who underwent gastrectomy and following radiation and chemotherapy.

Hou Gu Mi Xi is a dietary therapy form of Shen Ling Bai Zhu San, which removes atractylodes and platycodon grandiflorum (two herbs that could not be used as food) from Shen Ling Bai Zhu San, and adds perilla leaf for adapting a dietary therapy for a long-term use. Hou Gu Mi Xi uses the main formula of Shen Ling Bai Zhu San, so that it could theoretically maintain the treatment effects. Although the reliable health effects of Shen Ling Bai Zhu San has been proved in previous studies, Hou Gu Mi Xi is optimized in formula and its preparations changed from electuary to rice paste, so that its functional mechanism and efficacy may be different. Therefore, the investigators plan to perform a hospital-based randomized controlled trial, enroll patients from three hospitals in Nanchang City of Jiangxi Province in China, for assessing efficacy and safety of Hou Gu Mi Xi on digestive symptoms in patients with spleen qi deficiency and radical gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be diagnosed as gastric cancer by pathology and have received radical gastrectomy. They should finish the following radiotherapy and chemotherapy and the treatment for surgical complications (such as leak, stricture, and marginal ulcer).
* Patient should be constitution of spleen qi deficiency, that is, meet two primary symptoms of spleen deficiency + two primary symptoms of qi deficiency, or meet two primary symptoms of spleen deficiency + one primary symptoms of qi deficiency + one auxiliary symptoms, or meet one primary symptoms of spleen deficiency + one primary symptoms of qi deficiency + two secondary symptoms + one auxiliary symptoms as follow:

  1. Main symptoms of spleen deficiency: a) poor appetite; b) abnormal stool (loose, diarrhea); c) abdominal distention after meal or afternoon
  2. Main symptoms of qi deficiency: a) fatigue; b) tired mind and taciturnity
  3. Secondary symptoms: a) tastelessness, hypodipsia, like hot drink, polysialia; b) abdominal pain, as a result either patients like warm or press, or remit after meal, or occur when work; c) nausea and vomiting; d) fullness in stomach; e) abnormal bowel sounds; f) lean or puffiness; g) sallow complexion; h) powerless defecation weakness; i) edema
  4. Auxiliary symptoms: pale or swollen or teeth-printed tongue with thin and white fur
* Age ranges from 18 to 70 years; both male and female
* Patient should be in fair performance status, indicated by a score of Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Sign the informed consent

Exclusion Criteria:

* Stage IV gastric cancer according to the Japanese classification criteria [16]
* Impaired liver function (total bilirubin > 2 × upper limit of normal (ULN), alanine transaminase > 2 × ULN, or aspartate aminotransferase > 2 × ULN), kidney function (serum creatinine > 2 × ULN), or hematopoiesis (neutrophil counts < 0.5×109/L or, thrombocyte counts < 20×109/L or, absolute reticulocyte counts < 15×109/L)
* Obviously abnormal electrocardiogram
* Severe mental disorders
* Other severe diseases (e.g. multiple organ failure, HIV infection)
* Pregnant or breast-feeding women
* Allergic to the test sample
* Unwilling to provider personal information and sign the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in total scores of Spleen Qi Deficiency Symptoms Grading and Quantifying Scale (Units on a scale) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  Higher score indicates severer symptoms of Spleen Qi Deficiency. Units of measure (Units on a scale)

SECONDARY OUTCOMES:
Qualitative assessment of changes in total scores of SQD scale from baseline | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  1) completely remission: reduction in scores is ≥ 95% compared with baseline; 2) markedly effective: reduction in scores is 70% to 94% compared with baseline; 3) effective: reduction in scores is 30% to 69% compared with baseline; 4) not effective: reduction in scores is < 30% compared with baseline
Changes in scores of each item of SQD scale from baseline | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  1) Stomach distension*, 2) Abdominal distension*, 3) Fatigue and weakness*, 4) Tired mind and taciturnity*, 5) Inappetence*, 6) Stomach pain, 7) Stomach tightness, 8) Abdominal pain, 9) Acid reflux, 10) Belching, 11) Nausea and vomiting, 12) Abnormal stools, 13) Abnormal bowel sounds, 14) Powerless defecation, 15) Sallow complexion, 16) Tastelessness and hypodipsia, and 17) Face and limbs edema.
Changes from baseline in total scores of Short Form 36 (SF-36) (Units on a scale) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To assess quality of life
Changes from baseline in scores of subitems in Short Form 36 (SF-36) (Units on a scale) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  Physical Component Summary (PCS) and Mental Component Summary (MCS)
Changes from baseline in scores of Eastern Cooperative Oncology Group (ECOG) Performance Status (Units on a scale) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To assess performance status
Progression free survival (month) | From the first dose of intervention up to 104 weeks
  assessed by evidence of pathological examination, computed tomography and/or magnetic resonance imaging
Changes from baseline in systolic blood pressure (mmHg) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To determine whether the interventions improve systolic blood pressure
Changes from baseline in diastolic blood pressure (mmHg) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To determine whether the interventions improve diastolic blood pressure
Changes from baseline in body weight (kg) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To determine whether the interventions improve body weight
Changes from baseline in body mass index (kg/m2) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  To determine whether the interventions improve body mass index
Incidence of any adverse events | From the first dose of intervention up to 104 weeks
  abnormal results (indicated by more or less than 2 × normal reference interval) in the routine blood, urine, and stool tests, liver function tests (alanine transaminase [ALT], aspartate aminotransferase [AST], total bilirubin [TBIL], direct bilirubin [DBIL], indirect bilirubin [IBIL]), kidney function tests (serum creatinine [SCr] and urea nitrogen [BUN]), coagulation function (prothrombin time [PT], activated partial thromboplastin time [APTT], thrombin time [TT], fibrinogen [FIB]), and electrocardiogram as well as any other new-onset symptoms or diseases related or unrelated to the intervention
Incidence of severe adverse events | From the first dose of intervention up to 104 weeks
  AEs that lead to new or prolonged hospitalization, disability, admission to intensive care unit, life danger, and death
Incidence of drug-related adverse events | From the first dose of intervention up to 104 weeks
  This outcome is assessed by blinded clinicians in each research center
Incidence of withdrawn due to adverse events | From the first dose of intervention up to 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Zhu, Ph.D., Study Chair — Jiangxi University of Traditional Chinese Medicine
Locations (1):
- Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data.

REFERENCES:
- [Background] Oh SY, Lee HJ, Yang HK. Pylorus-Preserving Gastrectomy for Gastric Cancer. J Gastric Cancer. 2016 Jun;16(2):63-71. doi: 10.5230/jgc.2016.16.2.63. Epub 2016 Jun 24. PMID 27433390
- [Background] Yang L. Incidence and mortality of gastric cancer in China. World J Gastroenterol. 2006 Jan 7;12(1):17-20. doi: 10.3748/wjg.v12.i1.17. PMID 16440411
- [Background] Wu TH, Chen IC, Chen LC. Antacid effects of Chinese herbal prescriptions assessed by a modified artificial stomach model. World J Gastroenterol. 2010 Sep 21;16(35):4455-9. doi: 10.3748/wjg.v16.i35.4455. PMID 20845514
- [Background] Yin GY, Chen Y, Shen XJ, He XF, Zhang WN. Study on the pathophysiologic basis of classification of 'spleen' deficiency in chronic gastritis. Chin Med J (Engl). 2005 Mar 20;118(6):468-73. PMID 15788127
- [Background] Yin GY, Zhang WN, Shen XJ, He XF, Chen Y. Study on the pathological basis of classification of spleen deficiency in chronic gastritis. Chin Med J (Engl). 2004 Aug;117(8):1246-52. PMID 15361303
- [Derived] Zhou X, Yan DM, Zhu WF, Liu WJ, Nie HY, Xu S, Jiang YP, Zhang KH, Fu Y, Wan YY, Yu XY, Li H, Sun X, Chen XF. Efficacy and safety of Hou Gu Mi Xi in patients with spleen qi deficiency syndrome who underwent radical gastrectomy for gastric cancer: protocol for a multicenter, randomized, double-blind, placebo-controlled trial. Trials. 2019 Jun 10;20(1):343. doi: 10.1186/s13063-019-3429-x. PMID 31182140